CLINICAL TRIAL: NCT04851639
Title: The Wolverhampton Assessment Tool, a Step Towards Remote Monitoring of Patient-reported Wellbeing in the Context of Prostate Cancer
Brief Title: The Wolverhampton Assessment Tool, a Tool for Patient-reported Wellbeing in the Context of Prostate Cancer
Acronym: WATapp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wolverhampton (Other)
Collaborators: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Dr David Matheson, Principal Investigator, University of Wolverhampton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 284454
Record Dates: First submitted 2021-04-06; First posted 2021-04-20 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Advanced Prostate Carcinoma
Keywords: metastatic; quality of life; patient empowerment
MeSH Terms: conditions — Neoplasm Metastasis; Patient Participation

STUDY DESIGN:
Intervention Model Description: any patient with advanced or metastatic prostate cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proof of principle (Experimental): Proof of principle of the efficacy and utility of the WATapp
  Interventions: Other: Wolverhampton Assessment Tool

INTERVENTIONS:
Other: Wolverhampton Assessment Tool — a proxy means for assessing whether clinician intervention is required and to assess patient's lived quality of life

SUMMARY:
This is a study of the Wolverhampton Assessment Tool (WATapp), a five-item questionnaire for patients with advanced or metastatic prostate cancer to say how they feel normally in terms of pain, urinary frequency, eating, and tiredness. It is widely recognised that patient-reported outcomes give a measure of overall effect of clinicians' actions on patients and that they can be used to guide the management of the patient's condition.

WATapp is designed to reduce the need for the patient to attend hospital so much for routine follow-up consultations (an important aspect in light of COVID-19), to give the patient some sense of agency and control and to inform his clinician of just he feels he is coping with his treatment. Now the investigators want to find out just how the results from WATapp correspond to, for example, changes in the patient's PSA, testosterone or other blood results which are routinely measured; and to find out how patients and clinicians feel about using WATapp.

Men with advanced or metastatic prostate cancer will be eligible to take part in the study and participation is in addition to whatever treatment they are on. Clinicians who choose to offer WATapp to their patients will also be invited to take part and they will be asked to share with the researchers anonymised, linked patient data and scores from WATapp.

DETAILED DESCRIPTION:
It is widely recognised that patient-reported outcomes give a measure of overall effect of clinicians' actions on patients and that they can be used to guide the management of the patient's condition. They can also have an empowering effect as the patient may feel that they are agents, and not just subjects, in their treatment pathway. In the case of advanced and metastatic prostate cancer (i.e. cancer which has spread from the prostate to distant sites), the clinical means of assessing how the patient's disease is responding to treatment (radiological/magnetic scans) are somewhat imperfect as they do not take into account the impact on the patient's life and his response and reaction. Patient-reported outcomes, such as WATapp, allow a way to measure the impact of clinicians' actions on patients' lives. They offer an assessment of how well treatments are working and this is critical in the management of patients with advanced or metastatic prostate cancer. Failure to recognise how the patient responds to treatment can lead to effective treatment being stopped inappropriately; progression of the disease may not always be recognised; and the patient may have unnecessary side effects that go unchecked. Ignoring the patient-reported outcomes, such as WATapp, can reduce the opportunity to use alternative treatments. WATapp has been developed as an objective and reproducible clinical assessment tool by using questions from these validated clinical study tools:

The Functional Assessment of Cancer Therapy - Prostate; The Brief Pain Inventory; The Karnofsky Performance Scale

WATapp was refined with patient and clinician input to produced the present 5-item questionnaire.

This is a mixed-method study, incorporating both quantitative and qualitative elements. As such, it is both objective and subjective:

1. It is subjective in that, in using the WATapp, the patient selects his response to each question on the basis of how he feels normally
2. It is objective in that the tools to be used in the analysis of the quantitative data [i.e. statistical tests such as Mann Whitney-U, Spearman Rank Correlation etc.] are independent of the person using them
3. Determining clinically the patient's disease status employs objective measures such as PSA, size, distribution and type of metastasis, frequency of night-time urination etc. as well as the clinician's professional judgment which contains both objective and subjective elements
4. The researchers are not mirrors but rather prisms and hence the entire study from conception to analysis and report is a refraction of their experiences

Phase 1 The main outcome of the first phase will be to refine, as necessary, both the WATapp and the research instruments as well as to establish proof of principle of the clinical utility of WATapp. This will entail a full pilot of the WATapp in New Cross Hospital, Wolverhampton. Patients who agree to use the WATapp to self-monitor aspects of their health will be invited to consent to share with the researchers their anonymised data from it as well as linked, anonymised clinical data. The frequency of collection of data will be at the discretion of the clinician. Participating patients and clinicians will be invited to take part in a short, semi-structured interview on their experience of using WATapp. All patient data will be treated anonymously, and none linked back to the patient or to their clinician/s. Clinicians will be asked to record any reasons given by patients who decline to use the WATapp. Whether a patient chooses or not to use WATapp or chooses or not to take part in this study will have no bearing on their clinical care.

The clinical data sought on patients will include:

1. Age
2. Stage of cancer at diagnosis in terms of the primary tumour, and any presence of disease in lymph nodes and bones
3. Current stage of cancer in terms of the primary tumour, and any presence of disease in lymph nodes and bones
4. Level of PSA - prostate specific antigen, produced normally in the prostate but also produced in prostate cancer cells, testosterone and other blood results which are routinely measured
5. Any other illnesses the patient may have
6. Current and previous treatments

Phase 2 The second phase is to invite oncologists across the West Midlands of England, many of whom have already expressed an interest, to join the study and to send the researchers anonymised, linked patient data (as in Phase 1) and that from the WATapp.

ELIGIBILITY:
Inclusion Criteria:

* born male
* diagnosed with advanced or metastatic prostate cancer
* able to read and speak English

Exclusion Criteria:

* not born male
* not diagnosed with advanced or metastatic prostate cancer
* not able to read and speak English

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
WATapp as a proxy for patients' clinical status | up to 48 months
  The correlation between the patient's responses to WATapp and their clinical status as measured by routine bloods and clinician assessment.

CONTACTS AND LOCATIONS:
Overall Officials: David Matheson, PhD, Principal Investigator — University of Wolverhampton
Locations (1):
- Royal Wolverhampton Hospital NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The IPD plan is in development. It is expected that it will include
  * Study protocol
  * Information sheets and blank informed consent forms
  * Anonymised data from the study
  Sharing will be subject to application, guarantees as to usage, due recognition of source
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available once we have published our results and for two years thereafter.
Access Criteria: Data will be available to bona fide researchers with good reason such as conducting meta-analyses

DOCUMENTS (1):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04851639/Prot_000.pdf